CLINICAL TRIAL: NCT04012489
Title: Comparison Between Breath Stacking and Air Stacking on Respiratory Mechanics and Ventilatory Pattern in Tracheostomized Patients: Randomized Crossover Trial
Brief Title: Breath and Air Stacking on Respiratory Mechanics in Tracheostomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Institute of Higher Education of Censa (Other)
Responsible Party: Principal Investigator, Luciano Matos Chicayban, Laboratório de Pesquisa em Fisioterapia Pneumofuncional e Intensiva (LAPEFIPI), Brazilian Institute of Higher Education of Censa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Air and Breath Stacking
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Mechanical Ventilation; Lung Infection
Keywords: Physical Therapy Modalities; Respiratory Care Units; Respiratory Mechanics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath Stacking (Active Comparator): Breath stacking: patients were connected to a unidirectional valve coupled to artificial airway (tracheostomy), with bacteriological filter. The ventilator was coupled to the unidirectional valve to measure inspiratory volume mobilized in each cycle and a connection to adapt a manometer. The patient performed successive inspirations for a maximum period of 30 seconds or until unidirectional valve opening or volume increase was observed for 2 consecutive efforts. Ten cycles of the technique were performed, with an interval of 30 seconds.
  Interventions: Procedure: Breath Stacking
- Air Stacking (Experimental): Air stacking: the same system of monitoring and adaptation of the ventilometer and manometer was carried out. A manual resuscitator coupled to a unidirectional valve was used, both connected to the tracheostomy, with a filter interface. Slow and successive inspirations were performed through slow compression of the resuscitator until the maximum inspiratory pressure reached 40 cmH2O. Ten cycles of the technique were performed, with an interval of 30 seconds.
  Interventions: Procedure: Air Stacking

INTERVENTIONS:
Procedure: Breath Stacking — Patients were connected to a unidirectional valve coupled to artificial airway (tracheostomy), with bacteriological filter. The ventilator was coupled to the unidirectional valve to measure inspiratory volume mobilized in each cycle and a connection to adapt a manometer. The patient performed successive inspirations for a maximum period of 30 seconds or until unidirectional valve opening or volume increase was observed for 2 consecutive efforts. Ten cycles of the technique were performed, with an interval of 30 seconds.
  Arms: Breath Stacking
Procedure: Air Stacking — The same system of monitoring and adaptation of the ventilometer and manometer was carried out. A manual resuscitator coupled to a unidirectional valve was used, both connected to the tracheostomy, with a filter interface. Slow and successive inspirations were performed through slow compression of the resuscitator until the maximum inspiratory pressure reached 40 cmH2O. Ten cycles of the technique were performed, with an interval of 30 seconds.
  Arms: Air Stacking

SUMMARY:
The researchers hypothesized that the aid of the resuscitator by the technique Air Stacking increase lung volume, promoting increased lung compliance and improvement of the ventilatory pattern. In addition, Air Stacking does not depend on patient collaboration. The objective of this study was to compare the effects of breath stacking and air stacking techniques on respiratory mechanics and ventilatory pattern in patients admitted to the ICU

ELIGIBILITY:
Inclusion Criteria:

* Patients without mechanical ventilation for more than 72 hours
* Mucus hypersecretion (defined as the need for suctioning < 2-h intervals)

Exclusion Criteria:

* bronchospasm.
* Pleural effusion or pneumothorax undrained.
* Bronchopleural or tracheoesophageal fistula.
* Neuromuscular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Static compliance of respiratory system | Baseline (before) and immediately after Breath Stacking or Air Stacking
  Compliance was assessed through the occlusion maneuver at the end of inspiration, considering tidal volume, plateau pressure and PEEP. Three measurements were taken at each moment, the mean being used.
Total Resistance of respiratory system | Baseline (before) and immediately after Breath Stacking or Air Stacking
  The total resistance of the respiratory system was evaluated through the occlusion maneuver at the end of the inspiration, considering the resistive pressure, measured by the difference between the maximum plateau pressure. Three measurements were taken at each moment, the mean being used.

CONTACTS AND LOCATIONS:
Locations (1):
- Luciano M Chicayban, Campos dos Goytacazes, Rio de Janeiro, Brazil